CLINICAL TRIAL: NCT05904015
Title: A Prospective, Two Cohort, Multicenter Phase II Clinical Study of Envafolimab Combined With Concurrent Chemoradiotherapy and Immune Maintenance Therapy For Limited Stage Small Cell Lung Cancer
Brief Title: The Study of Envafolimab Combined With Concurrent Chemoradiotherapy In LS-SCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LVHUA WANG, professor of medicine, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT-LC03
Record Dates: First submitted 2023-04-30; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Lung Neoplasms
Keywords: Envafolimab/SCLC/Chemoradiotherapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated radiotherapy group (Experimental): Envafolimab: 300mg SC d1,Q3W,2 cycles Cisplatin/carboplatin: Cisplatin: 75 mg/m2 IV d1,Q3W ,2 cycles or Carboplatin:AUC=5/6 IV d1,Q3W,2cycles Etoposide: 100mg/m2 IV d1,Q3W ,2 cycles Radiotherapy: Provide a prescription dose of 45Gy at a 95% PTV dose, with a single split dose of 3Gy, once a day, 5 times a week, for a total of 15 times.
  Envafolimab maintenance: 300mg,SC, d1. Q3W, up to 2 years or until PD or intolerable.
  Interventions: Drug: Envafolimab combined with concurrent chemoradiotherapy (Hypofractionated radiotherapy)
- Conventional Radiotherapy (Experimental): Envafolimab: 300mg SC d1,Q3W,2 cycles Cisplatin/carboplatin:Cisplatin:75 mg/m2 IV d1,Q3W ,2 cycles or Carboplatin:AUC=5/6 IV d1,Q3W,2cycles Etoposide: 100mg/m2 IV d1,Q3W ,2 cycles Radiotherapy: Provide a prescription dose of 60Gy at a 95% PTV dose, with a single split dose of 2Gy, once per day, 5 times per week, for a total of 30 times Envafolimab maintenance: 300mg,SC, d1. Q3W, up to 2 years or until PD or intolerable.
  Interventions: Drug: Envafolimab combined with concurrent chemoradiotherapy (Conventional Radiotherapy)

INTERVENTIONS:
Drug: Envafolimab combined with concurrent chemoradiotherapy (Hypofractionated radiotherapy) — Envafolimab: 300mg SC d1,Q3W,2 cycles Cisplatin/carboplatin: Cisplatin: 75 mg/m2 IV d1,Q3W ,2 cycles or Carboplatin:AUC=5/6 IV d1,Q3W,2cycles Etoposide: 100mg/m2 IV d1,Q3W ,2 cycles Radiotherapy: Provide a prescription dose of 45Gy at a 95% PTV dose, with a single split dose of 3Gy, once a day, 5 times a week, for a total of 15 times.
  Envafolimab maintenance: 300mg,SC, d1. Q3W, up to 2 years or until PD or intolerable.
  Other Names: Hypofractionated Radiotherapy Group
  Arms: Hypofractionated radiotherapy group
Drug: Envafolimab combined with concurrent chemoradiotherapy (Conventional Radiotherapy) — Envafolimab: 300mg SC d1,Q3W,2 cycles Cisplatin/carboplatin:Cisplatin:75 mg/m2 IV d1,Q3W ,2 cycles or Carboplatin:AUC=5/6 IV d1,Q3W,2cycles Etoposide: 100mg/m2 IV d1,Q3W ,2 cycles Radiotherapy: Provide a prescription dose of 60Gy at a 95% PTV dose, with a single split dose of 2Gy, once per day, 5 times per week, for a total of 30 times.
  Envafolimab maintenance: 300mg,SC, d1. Q3W, up to 2 years or until PD or intolerable.
  Other Names: Conventional Radiotherapy Group
  Arms: Conventional Radiotherapy

SUMMARY:
To evaluate the efficacy and safety of envafolimab combined with concurrent chemoradiotherapy in limited stage small cell lung cancer.

DETAILED DESCRIPTION:
Envafolimab is the world's first subcutaneous injection of PD-L1 monoclonal antibody. Suitable for adult patients with advanced solid tumors with unresectable or metastatic microsatellite highly unstable (MSI-H) or mismatch repair gene defects (dMMR).

ELIGIBILITY:
Inclusion Criteria:

* The result of histopathological or cytological diagnosis is small cell lung cancer.
* Diagnosed as limited stage by imaging examination (lesion limited to half chest and one radiotherapy field, without malignant pleural or pericardial effusion); And at least one measurable lesion that meets the RECIST 1.1 standard.
* Have not received systematic treatment in the past, and initially underwent 2 cycles of etoposide+cisplatin/carboplatin induction therapy.
* Age 18-75 years old, male or non pregnant female.
* The expected survival period is>3 months.
* ECOG score 0-1.
* Weight>30 kilograms.
* All patients underwent chest CT, head MRI, abdominal CT or MRI, and whole body bone scan before treatment to clarify.
* Hematological indicators: white blood cell (WBC) count ≥ 4 * 109/L, absolute neutrophil count (ANC) ≥ 1.5 * 109/L, hemoglobin (Hb) level>100 g/L, platelet (Plt) count>100 * 109/L, serum creatinine (Cr) level<1.5 times the upper limit of normal value, serum alanine transaminase (AST) and glutamic transaminase (ALT) levels<2.5 times the upper limit of normal value, and serum bilirubin level ≤ 1.5 times the upper limit of normal value.
* The patient has signed an informed notice and is willing and able to comply with the visit, treatment plan, laboratory examination, and other research procedures of the research plan.

Exclusion Criteria:

* Patients with non-small cell lung cancer or mixed components of small cell lung cancer in histopathology.
* Patients with extensive stage small cell lung cancer (ES-SCLC).
* Merge malignant pleural effusion and pericardial effusion.
* Pregnant and lactating women.
* Merge patients with more severe underlying diseases.
* Patients who have previously been treated with inhibitors of immune regulatory points (CTLA-4, PD-1, PD-L1, etc.).
* Patients may require long-term use of immunosuppressive drugs or systemic or local use of corticosteroids with immunosuppressive doses for comorbidities.
* Patients with immunodeficiency disorders and a history of organ transplantation (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, nephritis, hyperthyroidism, hypothyroidism; vitiligo or childhood asthma. Patients who have completely relieved and do not require any intervention after adulthood can be included; asthma that requires medical intervention with bronchodilators cannot be included).
* Those whose laboratory test values during the screening period before enrollment do not meet relevant standards.
* Patients with significantly reduced heart, liver, lung, kidney, and bone marrow function.
* Serious and uncontrolled internal diseases and infections.
* Simultaneously using other investigational drugs or in other clinical trials.
* Refusal or inability to sign informed consent form for participation in the experiment.
* A history of allergies to etoposide, cisplatin, or any excipients.
* Researchers have determined that patients are not suitable to participate in the study and are unlikely to comply with the study procedures, limitations, and requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
2-year PFS rate | From date of randomization until the date of first documented progression or date of death from any cause up to 24 months.
  2-yaer progression-free survival rate

SECONDARY OUTCOMES:
ORR | From date of randomization until the date of first documented progression or date of death from any cause up to 24 months.
  Objective Response Rate
DCR | From date of randomization until the date of intolerance the toxicity or PD up to 24 months.
  Disease control rate
DOR | From date of randomization until the date of intolerance the toxicity or PD up to 24 months.
  Duration of response
OS | From date of randomization until the date of death(up to 24 months)
  Overall survival
Adverse event rate Adverse event rate Adverse event rate | From date of randomization until the date of toxicity or PD (up to 24 months)
  Number of participants with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: LvHua Wang, Doc, Study Chair — Cancer Hospital Chinese Academy of Medical Sciences,ShenZhen Cencer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Govindan R, Page N, Morgensztern D, Read W, Tierney R, Vlahiotis A, Spitznagel EL, Piccirillo J. Changing epidemiology of small-cell lung cancer in the United States over the last 30 years: analysis of the surveillance, epidemiologic, and end results database. J Clin Oncol. 2006 Oct 1;24(28):4539-44. doi: 10.1200/JCO.2005.04.4859. PMID 17008692
- [Background] Toh CK, Gao F, Lim WT, Leong SS, Fong KW, Yap SP, Hsu AA, Eng P, Koong HN, Thirugnanam A, Tan EH. Differences between small-cell lung cancer and non-small-cell lung cancer among tobacco smokers. Lung Cancer. 2007 May;56(2):161-6. doi: 10.1016/j.lungcan.2006.12.016. Epub 2007 Jan 31. PMID 17270313
- [Background] Sun JM, Choi YL, Ji JH, Ahn JS, Kim KM, Han J, Ahn MJ, Park K. Small-cell lung cancer detection in never-smokers: clinical characteristics and multigene mutation profiling using targeted next-generation sequencing. Ann Oncol. 2015 Jan;26(1):161-166. doi: 10.1093/annonc/mdu504. Epub 2014 Oct 29. PMID 25355724
- [Background] Sundstrom S, Bremnes RM, Kaasa S, Aasebo U, Hatlevoll R, Dahle R, Boye N, Wang M, Vigander T, Vilsvik J, Skovlund E, Hannisdal E, Aamdal S; Norwegian Lung Cancer Study Group. Cisplatin and etoposide regimen is superior to cyclophosphamide, epirubicin, and vincristine regimen in small-cell lung cancer: results from a randomized phase III trial with 5 years' follow-up. J Clin Oncol. 2002 Dec 15;20(24):4665-72. doi: 10.1200/JCO.2002.12.111. PMID 12488411